CLINICAL TRIAL: NCT01549951
Title: A Phase 2, Open-Label, Single-Arm, Multidose Study to Investigate the Effects of Orteronel on the QT/QTc Interval in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Study to Investigate the Effects of Orteronel on the QT/QTc Interval in Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C21012; 2012-000136-26 (EudraCT Number); U1111-1179-5656 (Registry Identifier: WHO)
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Cancer
Keywords: Metastatic castrate resistant prostate cancer, mCRPC, orteronel, TAK-700, Phase 2, QT, QTc
MeSH Terms: conditions — Prostatic Neoplasms | interventions — orteronel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Orteronel+Prednisone (Experimental)
  Interventions: Drug: Orteronel+Prednisone

INTERVENTIONS:
Drug: Orteronel+Prednisone — Orteronel 400-mg plus prednisone 5-mg will be administered BID orally continuously throughout the treatment cycle of the study.
  Other Names: TAK-700

SUMMARY:
The purpose of this phase 2, open-label, single-arm, multidose, multicenter study is to investigate the effects of Orteronel plus Prednisone on the QT/QTc interval in patients with Metastatic Castration-Resistant Prostrate Cancer

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written consent
* Screening PSA ≥ 2ng/ml
* Patients must have a diagnosis of mCRPC
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Prior surgical or medical castration with testosterone at screening < 50 ng/dL

Exclusion Criteria:

* Prior chemotherapy for prostate cancer within 6 months prior to screening. (Any prior therapy with cabazitaxel, mitoxantrone, or anthracyclines is exclusionary.)
* Documented central nervous system metastases
* Clinically significant heart disease
* Patients who have an abnormal 12-lead ECG result at screening including one or more of the following: QRS>110 ms, QTcF>480ms, PR interval>200 ms
* Patients who have a history of risk factors for TdP including unexplained syncope, known long QT syndrome, heart failure, angina, or clinically significant abnormal laboratory assessments

Please note that there are additional inclusion and exclusion criteria. The study center will determine if you meet all of the criteria.

Site personnel will explain the trial in detail and answer any question you may have if you do qualify for the study. You can then decide whether or not you wish to participate. If you do not qualify for the trial, site personnel will explain the reasons

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Pinnacle Oncology, Scottsdale, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 16 investigative sites in Canada, France, Greece, Ireland, Romania, and the United States from 29 May 2012 to 21 January 2015.
Pre-assignment Details: Male participants with a historical diagnosis of metastatic castration-resistant prostate cancer (mCRPC) were enrolled in this single arm study to receive orteronel 400 milligram (mg) along with prednisone 5 mg twice daily for 28 days in each treatment cycle.
Groups:
- Orteronel + Prednisone: Orteronel 400 mg, tablets, orally, twice daily along with prednisone 5 mg, tablets, orally, twice daily for 2 treatment cycles of 28 days each. Gonadotropin-releasing hormone analogue therapy was supplied as a commercially available dosage formulation.
Period: Overall Study
Arm/Group | Orteronel + Prednisone
Started | 50
Primary Reason Off Study Treatment | 50
Completed | 0
Not Completed | 50
Not completed — Adverse Event | 15
Not completed — Withdrawal by Subject | 2
Not completed — Unsatisfactory therapeutic response | 1
Not completed — Progressive disease | 29
Not completed — Symptomatic deterioration | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set was defined as all participants who received at least 1 dose of any study drug.
Arm/Group | Orteronel + Prednisone
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 22
Race/Ethnicity, Customized [Number; unit: participants]
  White | 27
  Black/African American | 3
  Not reported | 20
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 175.32 (7.521)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 87.63 (14.797)
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — ECOG assessed participant's performance status on 5point scale: 0=Fully active/able to carry on all pre-disease activities without restriction;1=restricted in physically strenuous activity,ambulatory/able to carry out light or sedentary work;2=ambulatory (greater than[>] 50 percent[%] of waking hours),capable of all self care,unable to carry out any work activities;3=capable of only limited selfcare,confined to bed/chair>50% of waking hours;4=completely disabled,cannot carry on any selfcare,totally confined to bed/chair;5=dead.Participants with performance status as 0 and 1 have been reported.
  participants
    0 | 38
    1 | 12
Histological classification [Number; unit: participants] — Carcinoma was classified as adenocarcinoma in situ (local), not otherwise specified (NOS) and adenocarcinoma, NOS.
  participants
    Adenocarcinoma in situ, NOS | 8
    Adenocarcinoma, NOS | 42
Time from initial prostate cancer diagnosis [Mean (Standard Deviation); unit: years] — Time from initial diagnosis was defined as (first dose date - initial diagnosis date + 1) / 365.25.
  years | 6.32 (5.325)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Change From Baseline in QTc Interval Based on the Fridericia Correction (QTcF) Method
Description: Triplicate 12-lead electrocardiogram (ECG) measurements (each recording separated by approximately 1 minute) were performed and average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR). Results of change in QTcF analyzed from 12-lead ECGs performed at each time point were averaged for analysis and a maximum across all post-dosing time points was used. Baseline is defined as the average of the triplicate 12-lead ECG measurements taken at the specified time prior to dosing.
Time Frame: Cycle 1 (28 day cycle), Day 1: pre-dose and at multiple timepoints (up to 6 hours) post-dose; Cycle 2 (28 day cycle), Day 1: pre-dose and at multiple timepoints (up to 6 hours) post-dose
Population: ECG analysis population was defined as all participants with at least 1 available baseline and at least 1 on-treatment ECG who received at least 1 dose of any study drug.
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | Orteronel + Prednisone
Number analyzed (Participants) | 43
millisecond (msec) | -1.4 (19.64)

2. Secondary Outcome: Maximum Change From Baseline in QTc Based on the Bazett Correction (QTcB) Method, PR, QRS and Uncorrected QT Interval
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 1 minutes) were performed and average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Bazette's formula (QTcB = QT divided by square root of RR). Results of change in QTcB, PR, QRS and uncorrected QT analyzed from 12-lead ECGs performed at each time point were averaged for analysis and a maximum across all post-dosing time points was used. Baseline is defined as the average of the triplicate 12-lead ECG measurements taken at the specified time prior to dosing.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Orteronel + Prednisone
Number analyzed (Participants) | 48
msec
  QTcB Interval (N=43) | 9.7 (22.61)
  PR Interval (N=48) | -4.2 (7.4)
  QRS Interval (N=48) | -1.0 (2.8)
  Uncorrected QT Interval (N=48) | -12.5 (17)

3. Secondary Outcome: Changes From Baseline in Heart Rate
Description: Triplicate 12-lead Electrocardiogram (ECG) measurements were performed and average was calculated. Supine heart rate was measured as beats per minute (bpm). Results of change in heart rate analyzed from 12-lead ECGs performed at each time point were averaged for analysis and a maximum across all post-dosing time points was used. Baseline is defined as the average of the triplicate 12-lead ECG measurements taken at the specified time prior to dosing.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Orteronel + Prednisone
Number analyzed (Participants) | 48
bpm | 5.7 (8.0)

4. Secondary Outcome: Number of Participants Reporting Change From Baseline in ECG Morphology
Description: Participants with incidence of ECG morphology abnormalities were observed. Types of abnormalities included appearance of abnormal U waves, T waves inversion, elevation of ST segment, depression of ST segment, second or third degree heart block, right or left bundle branch block, atrial fibrillation/flutter, and myocardial infarction. New morphological changes were observed in abnormal U waves, depression of ST segment, and T waves inversion. Here, 'new' refers to change not present at baseline, ie, at any evaluation predose, and only seen postbaseline. Results of change in ECG morphology analyzed from 12-lead ECGs at each time point were averaged for analysis and a maximum across all post-dosing time points was used. Baseline is defined as the average of the triplicate 12-lead ECG measurements taken at the specified time prior to dosing.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participant
Arm/Group | Orteronel + Prednisone
Number analyzed (Participants) | 48
participant
  Abnormal U waves | 1
  ST segment depression | 8
  T-wave inversion | 3

5. Secondary Outcome: Correlation Between the QTcF Change From Baseline and Plasma Concentrations of Orteronel
Description: Coefficient of correlation was measured using linear mixed effects model for the association between two variables; change from baseline versus the plasma concentration. Participant's effects on the intercept and plasma concentration slope were included in the model as random effects terms. Plasma concentrations were re scaled for model convergence. Average results at each time point were analyzed and a maximum across all post-dosing time points was used. Baseline is defined as the average of the triplicate 12-lead ECG measurements taken at the specified time prior to dosing.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: correlation coefficient
Arm/Group | Orteronel + Prednisone
Number analyzed (Participants) | 48
correlation coefficient | -0.002603 (0.001053)

6. Secondary Outcome: AUC(0-6): Area Under the Plasma Concentration-Time Curve From Time 0 to 6 Hours Postdose for Orteronel and M-I Metabolite
Description: AUC(0-6) is measure of area under the curve over the dosing interval (tau) (AUC(0-tau]), where tau is the length of the dosing interval - 6 hours in this study). Average results at each time point were analyzed and a maximum across all post-dosing time points was used. Baseline is defined as the average of the triplicate 12-lead ECG measurements taken at the specified time prior to dosing.
Time Frame: as for outcome 1
Population: Pharmacokinetic (PK) population was defined as all participants who had sufficient dosing data and plasma concentration-time data to permit calculations of PK parameters.
Measure: Mean (Standard Deviation); unit: nanogram hours per milliliter (ng*hr/mL)
Arm/Group | Orteronel + Prednisone
Number analyzed (Participants) | 50
nanogram hours per milliliter (ng*hr/mL)
  Cycle 1 Day 1 (n=50) | 7570.4 (3673.31)
  Cycle 2 Day 1 (n=44) | 12971.6 (6071.18)

7. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Orteronel and M-I Metabolite
Description: Tmax: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax. Average results at each time point were analyzed and a maximum across all post-dosing time points was used. Baseline is defined as the average of the triplicate 12-lead ECG measurements taken at the specified time prior to dosing.
Time Frame: as for outcome 1
Population: PK population was defined as all participants who had sufficient dosing data and plasma concentration-time data to permit calculations of PK parameters.
Measure: Median (Full Range); unit: hours
Arm/Group | Orteronel + Prednisone
Number analyzed (Participants) | 50
hours
  Orteronel: Cycle 1 Day 1 (n=50) | 2.0 [1.0 to 5.0]
  Orteronel: Cycle 2 Day 1 (n=44) | 1.6 [0.5 to 6.0]
  M-I metabolite: Cycle 1 Day 1 (n=50) | 4.5 [1.5 to 6.2]
  M-I metabolite: Cycle 2 Day 1 (n=44) | 3.0 [0.0 to 6.1]

8. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Orteronel and M-I Metabolite
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve. Average results at each time point were analyzed and a maximum across all post-dosing time points was used. Baseline is defined as the average of the triplicate 12-lead ECG measurements taken at the specified time prior to dosing.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Orteronel + Prednisone
Number analyzed (Participants) | 50
nanogram per milliliter (ng/mL)
  Orteronel: Cycle 1 Day 1 (n=50) | 1904.0 (1000.98)
  Orteronel: Cycle 2 Day 1 (n=44) | 3017.9 (1512.33)
  M-I metabolite: Cycle 1 Day 1 (n=50) | 263.5 (161.22)
  M-I metabolite: Cycle 2 Day 1 (n=44) | 597.5 (333.39)

9. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Baseline up to 30 days after last dose of study drug (Day 86)
Population: Safety analysis set was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Orteronel + Prednisone
Number analyzed (Participants) | 50
participants | 48

10. Secondary Outcome: Number of Participants Reporting Clinically Significant Abnormalities in Laboratory Values
Description: The number of participants with any clinically significant abnormalities in safety laboratory values collected throughout study.
Time Frame: Baseline up to 30 days after last dose of study drug (Day 86)
Population: Safety analysis set was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Orteronel + Prednisone
Number analyzed (Participants) | 50
participants | 5

11. Secondary Outcome: Number of Participants Reporting Clinically Significant Abnormalities in Vital Signs
Description: The number of participants with any clinically significant abnormalities in vital signs collected throughout study. Vital signs included body temperature (oral), sitting blood pressure (after the participant has rested for at least 5 minutes), and pulse (bpm).
Time Frame: Baseline up to 30 days after last dose of study drug (Day 86)
Population: Safety analysis set was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Orteronel + Prednisone
Number analyzed (Participants) | 50
participants | 0

12. Secondary Outcome: Number of Participants Reporting Clinically Significant Abnormalities in Physical Findings
Description: Physical examination consists of examinations of the following body systems: (1) eyes; (2) ears, nose, throat; (3) cardiovascular system; (4) respiratory system; (5) gastrointestinal system; (6) dermatologic system; (7) extremities; (8) musculoskeletal system; (9) nervous system; (10) lymph nodes; and (11) physical examinations other than body systems described in (1) to (10).
Time Frame: Baseline up to 30 days after last dose of study drug (Day 86)
Population: Safety analysis set was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Orteronel + Prednisone
Number analyzed (Participants) | 50
participants | 0

13. Secondary Outcome: Number of Participants Reporting Clinically Significant Abnormalities in ECG
Description: The number of participants who reported clinically significant abnormalities in ECG were measured throughout study. ECGs were performed after the participant had been supine for at least 10 minutes.
Time Frame: Baseline up to 30 days after last dose of study drug (Day 86)
Population: Safety analysis set was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Orteronel + Prednisone
Number analyzed (Participants) | 50
participants | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 30 days after the last dose of double-blind study drug (Day 86).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Orteronel + Prednisone
Serious Adverse Events (participants affected / at risk) | 17/50
Other Adverse Events (participants affected / at risk) | 48/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Orteronel + Prednisone (N=50)
Pumonary embolism (Respiratory, thoracic and mediastinal disorders) | 5
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Proctitis haemorrhagic (Gastrointestinal disorders) | 1
Bacteraemia (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia pseudomonal (Infections and infestations) | 1
Lung infection pseudomonal (Infections and infestations) | 0
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Angina pectoris (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Deep vein thrombosis (Vascular disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Blood glucose increased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Cerebrovascular disorder (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Orteronel + Prednisone (N=50)
Constipation (Gastrointestinal disorders) | 18
Nausea (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5
Fatigue (General disorders) | 12
Asthenia (General disorders) | 11
Decreased appetite (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 5
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Weight decreased (Investigations) | 9
Gamma-glutamyltransferase increased (Investigations) | 5
Rash macular (Skin and subcutaneous tissue disorders) | 4
Depression (Psychiatric disorders) | 6
Hot flush (Vascular disorders) | 7
Anaemia (Blood and lymphatic system disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Dysgeusia (Nervous system disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Alanine aminotransferase increased (Investigations) | 3
Blood lactate dehydrogenase increased (Investigations) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Dry mouth (Gastrointestinal disorders) | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3
Fall (Injury, poisoning and procedural complications) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Oedema peripheral (General disorders) | 3
Paraesthesia (Nervous system disorders) | 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3
Blood alkaline phosphatase increased (Investigations) | 4
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.